CLINICAL TRIAL: NCT03541889
Title: Multi-institutional Prospective Pilot Research of Imaging and Blood Biomarker EValuation of Engraftment After ALlogeneic Hematopoietic Stem Cell Transplantation
Brief Title: REVEAL Biomarkers of Engraftment After Alternative Donor HSCT
Acronym: REVEAL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Emory University (Other); University of Michigan (Other); University Hospitals Cleveland Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OU-SCC-REVEAL; 5R01HL146668-04 (NIH)
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Primary Graft Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cord and haplo imaging cohort (Experimental): For all pediatric and adult patients undergoing cord blood HSCT, FLT PET/CT imaging will occur one day prior to HSCT and on days 9 and 28 after HSCT. For recipients of haplo-HSCT, FLT PET/CT imaging will occur one day prior to HSCT and on days 5 and 28 after HSCT.
  Interventions: Drug: FLT imaging and TK1 blood measurements
- Nonengrafted cohort (Experimental): Pediatric and adult patients who have not engrafted by day 24 after cord or haplo-identical HSCT will undergo a single FLT PET/CT image within one week to determine if this scan can identify graft failure versus delayed engraftment.
  Interventions: Drug: FLT imaging and TK1 blood measurements

INTERVENTIONS:
Drug: FLT imaging and TK1 blood measurements — F18 labeled thymidine PET/CT scans will be performed. Serum measurements of TK1 will be obtained.

SUMMARY:
The purpose of this study is to find new tests that could help determine if the newly infused bone marrow cells are growing well after bone marrow transplantation or if new bone marrow cells are needed. The Investigator will use FLT imaging, an investigational imaging test, and collect blood samples to investigate whether the cells are growing well.

DETAILED DESCRIPTION:
This is a prospective pilot study with primary aim of determining whether investigational FLT imaging can detect and distinguish nonengraftment from delayed engraftment after HSCT in populations at highest risk for graft failure. The investigator will enroll up to 56 patients to achieve 50 evaluable patients undergoing hematopoietic cell transplantation on this trial [5 pediatric and adult recipients of cord blood stem cells (Arm A1), 15 pediatric and adult recipients of myeloablative haplo-identical HSCT (Arm A2), 10 pediatric and adult recipients of reduced intensity haplo-identical HSCT (Arm A3), and 20 recipients of these two stem cell sources who have not engrafted by day 28 (Arm B)]. Should a patient be unable to undergo FLT evaluation after enrollment or relapse in the first 30 days, the patient will be replaced. The planned length of this trial is 7 years and it will be conducted at 4 centers enrolling participants: Emory/Children's Healthcare of Atlanta, University of Oklahoma, University of Michigan, and University Hospitals of Cleveland.

For all pediatric and adult patients undergoing cord blood HSCT, FLT imaging will occur one day prior to HSCT and on days 9 and 28 after HSCT (Arm A1). For recipients of haplo-HSCT, FLT PET/CT imaging will occur one day prior to HSCT and on days 5 or 9 and 28 after HSCT (Arm A2 and A3). Pediatric and adult patients who have not engrafted by day 20 after cord or haplo-identical HSCT will undergo a single FLT image within one week to determine if this scan can identify graft failure versus delayed engraftment (Arm B). All patients will undergo serial peripheral blood evaluation for blood biomarker analysis, including thymidine kinase-1 (TK1). Study endpoints include: 1) detection of nonengraftment with FLT and TK1, 2) development of a model that predicts nonengraftment versus delayed engraftment using FLT and TK1, 3) sensitivity of individual biomarkers to distinguish between graft failure and delayed engraftment, and 4) biology of cord blood and haplo-HSCT engraftment.

For all pediatric and adult patients undergoing cord blood HSCT, three FLT images will be taken: first, one day prior to HSCT and second and third, on days 9 and 28 after HSCT. For recipients of haplo-HSCT, the FLT images will be taken one day prior to HSCT and then on days 5 and 28 after HSCT. Pediatric and adult patients who have not engrafted by day 24 after cord or haplo-identical HSCT will undergo a single FLT PET/CT image within one week, to determine if this scan can identify graft failure versus delayed engraftment. Blood samples will also be collected from all patients for blood biomarker analysis, including thymidine kinase-1 (TK1). Each patient will be in this study for one year.

ELIGIBILITY:
Inclusion Criteria:

General

* Ability to undergo 18F FLT imaging without sedation
* Patients > 4 years of age and less than 80 years of age at highest risk for graft failure: cord blood HSCT, haplo HSCT, or lack of engraftment by day 28.
* Diagnosed with a condition for which hematopoietic stem cell transplant (HSCT) is standard of care and HSCT is planned (Arm A) or occurred (Arm B)
* In morphologic remission prior to HSCT
* Patient or guardian able to give informed consent
* Investigational therapies within past 28 days or planned on protocol are pre-approved by the PI or Site PI
* Karnofsky or Lansky performance status > 60%

Arm A

* A1 Cord blood recipients: Absence of donor specific antibodies to cord HLA
* Haplo-identical recipients: ≥ 5/10 and < 7/8 allele mismatch donor
* A2- myeloablative Haplo-identical transplant is planned
* A3- reduced intensity Haplo-identical transplant is planned (non-myeloablative is excluded)
* A1- myeloablative or reduced intensity transplant is planned (non-myeloablative is excluded)
* Diagnosed with a condition for which hematopoietic stem cell transplant (HSCT) is standard of care and HSCT is planned
* Total bilirubin < 2.5 mg/dL (unless documented Gilbert's syndrome) and transaminases (ALT and AST) < 5 x the upper limit of normal
* Creatinine clearance or GFR > 60 ml/min/1.73 m2. (performed pre-HSCT)
* FEV1 > 80% pre or post-bronchiolator whichever is higher and DLCO Adj > 70% (performed pre-HSCT if age appropriate) and Sa02 > 94% on room air
* Ejection fraction > 50% (performed pre-HSCT)

Arm B

• Non-engraftment recipients of HCT with any donor source (related or unrelated): primary graft failure as defined by ANC not > 500 for 3 consecutive days and at least 20 days after HSCT.

Inclusion Criteria - Donors

* 1-2 cords and >.4/6 match to recipient for each (as per current National Marrow Donor guidelines), with a dose >2 x 10e6 CD34 cells/kg for each cord OR > 5/10 and <7/8 allele mismatch related donor
* Institutional guidelines met for donor suitability

Exclusion Criteria:

* History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent
* Clinically significant systemic illness with manifestations of significant organ dysfunction which, in the judgment of the PI, or Co-I, would render the patient unlikely to tolerate the protocol therapy or complete the study
* Presence of active malignancy from an organ system other than hematopoietic
* Pregnant or lactating females
* Patients who are unable or unwilling to use effective form (s) of contraception during the course of the study
* Prior history of fluorothymidine allergy or intolerance
* Decline enrolment on CIBMTR research protocol

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
FLT SUV identifies graft failure | 24-28 days
  To calculate if SUV > 1.2 identifies subclinical engraftment using FLT PET/CT imaging for recipients of cord and haplo-HSCT who have not engrafted within 24 days of HSCT.

SECONDARY OUTCOMES:
Map subclinical engraftment in alternative donor HSCT | Day -1 to Day 28 after HSCT
  Use SUV increase in particular medullary spaces to identify the first site of marrow settling after HSCT in alternative donor HSCT
TK1 serum levels identify graft failure | 24-28 days
  Calculate if TK1 level increases correlate with clinical engraftment
Number of patients with CTCAE version 5 events exceeding grade 3 that are possibly, probably, or definitely attributed to the FLT imaging | Day -1 to Day 28 after HSCT
  Safety of FLT in alternative donor HSCT - Calculate the number of patients with CTCAE version 5 events exceeding grade 3 that are possibly, probably, or definitely attributed to the FLT imaging
Other cytokine and chemokine markers of graft failure | 24-28 days
  Explore other cellular, cytokine, and chemokine markers of subclinical engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Williams, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University Hospital of Cleveland UH Seidman Cancer Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No